CLINICAL TRIAL: NCT06630637
Title: Intermittent Fasting Monitoring for Human Optimization Utilizing Wearable Technology: an N-of-1 Prospective Study
Brief Title: Monitoring Intermittent Fasting for Human Optimization Using Wearable Technology: An N-of-1 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Digital Medicine (WisDM) (Other)
Responsible Party: Principal Investigator, Dean Ho, Director of the N.1 Institute for Health, The N.1 Institute for Health (N.1)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HO_prospective
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Intermittent Fasting; Healthy; Digital Health
Keywords: Continuous Glucose Monitoring (CGM); Intermittent Fasting (IF); Ketone Measurement; Wearable Technology; Exercise Routines; Heat/Cold Interventions; Diet and Supplements; Human Optimization; N-of-1; Single Participant; Personalized Health; Digital Health; Sensors
MeSH Terms: conditions — Intermittent Fasting; Ketosis | interventions — Continuous Glucose Monitoring; Hematologic Tests; Occult Blood; Cold Temperature; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: This is an N-of-1 trial involving a single participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized Health Intervention Arm (Experimental): This arm involves the the single participant following a personalized regimen that includes intermittent fasting, exercise routines, heat/cold interventions, diet modifications, and supplementation. The participant will engage in continuous monitoring of metabolic changes using wearable technology, continuous glucose monitoring, and ketone measurements, along with blood, saliva, and stool lab tests. The goal is to assess the effects of these interventions on metabolic health and overall well-being, identifying potential trends and correlations throughout the study period.
  Interventions: Behavioral: Glucose-Ketone Index (GKI) monitoring; Behavioral: Continuous Glucose Monitoring (CGM); Other: Digital dynamometer; Device: Wearables; Diagnostic Test: Blood tests; Diagnostic Test: Stool tests; Diagnostic Test: Saliva tests; Behavioral: Fitness intervention; Behavioral: Cold & heat intervention; Device: Airofit; Behavioral: 18h fasting; Behavioral: 48h fasting; Behavioral: Three meal phase; Behavioral: Mediterranean-inspired diet; Dietary Supplement: Supplements; Behavioral: Generative AI; Other: Interviews

INTERVENTIONS:
Behavioral: Glucose-Ketone Index (GKI) monitoring — Ketone and blood glucose monitoring with Abbott Optium Neo up to 10 times per day to observe GKI dynamics for gamification of adherence.
Behavioral: Continuous Glucose Monitoring (CGM) — Monitoring with an Abbott Freestyle Libre to observe glucose dynamics for gamification of adherence.
Other: Digital dynamometer — Grip strength measurements, right and left hand, up to 20 readings per day per hand.
Device: Wearables — All Apple Watch 9 and Whoop data daily [heart rate variability (HRV), resting heart rate, cardio recovery, sleep duration, composition (stages of sleep) and analogous scores, potential maximum rate of oxygen consumption attainable during physical exertion (VO2 max), basal metabolic rate and potential respiratory rate].
Diagnostic Test: Blood tests — Pre- and Post-fast (48h) testing of lipid panel, ApoB, ApoA1, CRP, interleukin panel, omega 3:6 ratio, and autophagy analysis. Potential CBC, renal and liver panels to be taken where appropriate.
Diagnostic Test: Stool tests — 15 g of stool will be collected from the subject pre- and post-fast for microbiome assessment and pre- and post- the first week (the "three meal phase"). After the first week, the maximum number of tests is four per month (maximum of two fasts, with a pre- and post-fast test for each fast).
Diagnostic Test: Saliva tests — Saliva samples will be collected from the subject pre- and post-fast for microbiome assessment. Maximum number of tests is four per month (maximum of two fasts, with a pre- and post-fast test for each fast).
Behavioral: Fitness intervention — 90 minutes of strength and/or cardiovascular training for a minimum of 5 days per week.
Behavioral: Cold & heat intervention — Cold plunge: at least 3 days per week, 2 sessions of maximum 5 minutes each (minimum 2 minutes between sessions) at a minimum of 6 degrees Celsius. Potential inclusion of GKI measurements before and after plunge.
  Heat Therapy: maximum of 2 sessions of 20 minutes each of dry sauna blanket (minimum 5 minutes break between sessions) following the cold plunge intervention.
Device: Airofit — Airofit is a smart breathing training device designed to improve respiratory strength and efficiency. It is used for enhancing sport performance, well-being, and overall health. The device works by providing adjustable resistance to breathing muscles.
  5-10 minutes of daily use.
Behavioral: 18h fasting — Minimum of 18 hours fasting per day, with feeding window to occur between 5pm-8pm or 12pm-3pm. The fasting procedures will occur only after the Three Meal Phase.
Behavioral: 48h fasting — 48h fasting maximum twice monthly, at least one week apart. Multivitamin and electrolytes with water, and black coffee or tea (0-calorie drinks) will be consumed.The fasting procedures will occur the Three Meal Phase.
Behavioral: Three meal phase — During the first week of the study, the participant will follow a regime of three meals per day.
Behavioral: Mediterranean-inspired diet — Regimen of Mediterranean-inspired nutrition comprised of Olive Oil, Olives, Leafy Green Vegetables, Lean Protein (Beef, Chicken, Lamb, Pork, Duck, Salmon, Tuna), Chia Seeds, Pecans, Macadamia, Pumpkin Seeds, Walnuts, Greek Yogurt, Salt, Pepper, Paprika, Cumin, Garlic powder, onion powder; Fruit: Blueberry, Grapefruit; Carbohydrates: Rolled Oats; Hydration: Water, Black Coffee, Black Tea, Coke Zero and 100 Zero sparingly, Ultima electrolytes.
  Photographs of meals will be taken to create a visual record of the diet followed. Photographs of the devices will be taken to create a visual record of the blood glucose and ketone concentration results.
Dietary Supplement: Supplements — Multivitamin (Centrum), Vitamin D (Up to 2000 IU per day), Creatine (Up to 2000mg), Fisetin (1 pill), Omega-3 (1 tablet), Turmeric, Pre-Probiotic, Blueberry Extract, Holy Basil Extract.
Behavioral: Generative AI — Feeding ketone data, glucose data (from finger prick and/or CGM), any/all Apple Watch Data, and dietary images into a generative AI platform to convert data into images using any selected prompts, with the intent of the images serving as immediate, visual readouts as a function of activity and/or inactivity.
Other: Interviews — Three interviews, of 30-60 minutes each one, at baseline, end of three meal phase and end of study, to gain insights into the participant's experience. Exploration of daily routines including diet, exercise and the use of technology and aspects of a healthy lifestyle.

SUMMARY:
There is a growing interest in personalized health strategies, including diet, exercise, and fasting regimens, to enhance metabolic fitness. Recent research indicates that intermittent fasting (IF) is useful not only for weight management, but also for energy production and improvement of metabolic well-being.

IF can potentially reduce systemic inflammation and help to prevent chronic diseases. IF research can also help athletes sustain performance during fasting periods. This prospective study aims to investigate the effects of a human optimization program on an individual's metabolic health and overall well-being.

This research examines the correlations between continuous glucose monitoring, ketone measurement, exercise routines, heat/cold interventions, diet, supplements and intermittent fasting patterns. The study involves a single participant -the principal investigator- who will adhere to a personalized regimen involving wearable monitoring of metabolic changes, training and intermittent fasting. This research seeks to understand the potential relationships between these factors, contributing to the emerging knowledge on individualized health optimization.

ELIGIBILITY:
Inclusion Criteria:

* The principal investigator is the sole participant in this N-of-1 trial: a healthy individual with no chronic diseases or conditions affecting metabolic health.

Exclusion Criteria:

* The principal investigator is the sole participant in this N-of-1 trial.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Metabolic biomarker analysis: total cholesterol levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of total cholesterol: milligrams per deciliter (mg/dL)
Metabolic biomarker analysis: low density lipoprotein (LDL) cholesterol levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of LDL cholesterol: milligrams per deciliter (mg/dL)
Metabolic biomarker analysis: high density lipoprotein (HDL) cholesterol levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of HDL cholesterol: milligrams per deciliter (mg/dL)
Metabolic biomarker analysis: triglycerides levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of triglycerides: milligrams per deciliter (mg/dL)
Metabolic biomarker analysis: apolipoprotein B (ApoB) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of apolipoprotein B (ApoB): milligrams per deciliter (mg/dL)
Metabolic biomarker analysis: apolipoprotein A1 (ApoA1) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of apolipoprotein A1 (ApoA1): milligrams per deciliter (mg/dL)
Metabolic biomarker analysis: C reactive protein (CRP) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of C reactive protein (CRP): milligrams per liter (mg/L)
Metabolic biomarker analysis: interleukin 1β (IL- 1β) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of IL- 1β: picograms per milliliter (pg/mL)
Metabolic biomarker analysis: interleukin 6 (IL- 6) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of IL-6: picograms per milliliter (pg/mL)
Metabolic biomarker analysis: interleukin 8 (IL- 8) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of IL-8: picograms per milliliter (pg/mL)
Metabolic biomarker analysis: interleukin 10 (IL- 10) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of IL-10: picograms per milliliter (pg/mL)
Metabolic biomarker analysis: interleukin 12 (IL- 12) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of IL-12: picograms per milliliter (pg/mL)
Metabolic biomarker analysis: interleukin 17 (IL- 17) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of IL-17: picograms per milliliter (pg/mL)
Metabolic biomarker analysis: omega 3:6 ratio | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of omega 3:6 ratio (no specific units)
Metabolic biomarker analysis: Microtubule-associated protein 1A/1B-light chain 3 (LC3) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of autophagy biomarker LC3: Nanograms per milliliter (ng/mL)
Metabolic biomarker analysis: Sequestosome 1 (p62/SQSTM1) levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of autophagy biomarker p62/SQSTM1: Nanograms per milliliter (ng/mL)
Metabolic biomarker analysis: Beclin-1 levels | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood testing of autophagy biomarker Beclin-1: Nanograms per milliliter (ng/mL)
Metabolic biomarker analysis: Red Blood Cells (RBCs) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Red Blood Cells (RBCs): Million cells per microliter (million/µL)
Metabolic biomarker analysis: White Blood Cells (WBCs) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  White Blood Cells (WBCs): Thousand cells per microliter (thousand/µL)
Metabolic biomarker analysis: Hemoglobin (Hb) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Hemoglobin (Hb): Grams per deciliter (g/dL)
Metabolic biomarker analysis: Hematocrit (Hct) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Hematocrit (Hct): Percentage (%)
Metabolic biomarker analysis: Platelets (PLT) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Platelets (PLT): Thousand cells per microliter (thousand/µL)
Metabolic biomarker analysis: Blood Urea Nitrogen (BUN) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Blood Urea Nitrogen (BUN): Milligrams per deciliter (mg/dL)
Metabolic biomarker analysis: Creatinine | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Creatinine: Milligrams per deciliter (mg/dL) Estimated Glomerular Filtration Rate (eGFR): Milliliters per minute per 1.73 square meters (mL/min/1.73m²) Sodium: Milliequivalents per liter (mEq/L) Potassium: Milliequivalents per liter (mEq/L) Chloride: Milliequivalents per liter (mEq/L)
Metabolic biomarker analysis: Estimated Glomerular Filtration Rate (eGFR) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Estimated Glomerular Filtration Rate (eGFR): Milliliters per minute per 1.73 square meters (mL/min/1.73m²)
Metabolic biomarker analysis: Sodium | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Sodium: Milliequivalents per liter (mEq/L)
Metabolic biomarker analysis: Potassium | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Potassium: Milliequivalents per liter (mEq/L)
Metabolic biomarker analysis: Chloride | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Chloride: Milliequivalents per liter (mEq/L)
Metabolic biomarker analysis: Alanine Aminotransferase (ALT) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Alanine Aminotransferase (ALT): Units per liter (U/L)
Metabolic biomarker analysis: Aspartate Aminotransferase (AST) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Aspartate Aminotransferase (AST): Units per liter (U/L) Alkaline Phosphatase (ALP): Units per liter (U/L) Total Bilirubin: Milligrams per deciliter (mg/dL) Albumin: Grams per deciliter (g/dL)
Metabolic biomarker analysis: Alkaline Phosphatase (ALP) | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Alkaline Phosphatase (ALP): Units per liter (U/L)
Metabolic biomarker analysis: Total Bilirubin | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Total Bilirubin: Milligrams per deciliter (mg/dL)
Metabolic biomarker analysis: Albumin | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Albumin: Grams per deciliter (g/dL)
Microbial diversity | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Stool/saliva analysis of microbial diversity: Shannon diversity index (no specific units)
Taxonomic abundance | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Stool/saliva analysis of taxonomic abundance: reads per million (RPM)
Concentrations of metabolites | Pre and post 48 hour fasts (2 fasts per month for 12 months)
  Stool/saliva analysis of concentrations of metabolites: Micromoles per liter (µmol/L)
Glycemic and ketone monitoring for adherence assessment | 10 times per day for up to 12 months
  Glucose-Ketone Index (GKI): A calculated value derived from dividing the blood glucose level (in mmol/L) by the ketone level (in mmol/L).
Wearable health metrics analysis for physiological monitoring | Daily for up to 12 months
  Apple Watch 9 and Whoop data [heart rate variability (HRV), resting heart rate, cardio recovery, sleep duration, composition (stages of sleep) and analogous scores, potential maximum rate of oxygen consumption attainable during physical exertion (VO2 max), basal metabolic rate and potential respiratory rate].
Artificial intelligence (AI)-enhanced visual data representation for activity monitoring | Once a month for up to 12 months
  Feeding ketone data, glucose data, any/all wearable data, and dietary images into a generative AI platform to convert data into images using any selected prompts, with the intent of the images serving as immediate, visual readouts as a function of activity and/or inactivity.

OTHER OUTCOMES:
Qualitative assessment of participant experience | Day one, day 8, at study completion (12 months)
  This outcome involves conducting interviews with the participant to gather qualitative data on the experiences, challenges, and adherence related to the dietary and exercise interventions throughout the study. The interviews aim to provide insights into the participant's perceptions of the interventions, their effects on metabolic health and overall well-being, and any adjustments needed for optimal adherence and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Ho, PhD, Principal Investigator — The Institute for Digital Medicine (WisDM)
Locations (1):
- The Institute for Digital Medicine (WisDM), Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mandal S, Simmons N, Awan S, Chamari K, Ahmed I. Intermittent fasting: eating by the clock for health and exercise performance. BMJ Open Sport Exerc Med. 2022 Jan 7;8(1):e001206. doi: 10.1136/bmjsem-2021-001206. eCollection 2022. PMID 35070352
- [Background] Patterson RE, Sears DD. Metabolic Effects of Intermittent Fasting. Annu Rev Nutr. 2017 Aug 21;37:371-393. doi: 10.1146/annurev-nutr-071816-064634. Epub 2017 Jul 17. PMID 28715993
- [Background] Levy E, Chu T. Intermittent Fasting and Its Effects on Athletic Performance: A Review. Curr Sports Med Rep. 2019 Jul;18(7):266-269. doi: 10.1249/JSR.0000000000000614. PMID 31283627
- [Background] Tinsley GM, La Bounty PM. Effects of intermittent fasting on body composition and clinical health markers in humans. Nutr Rev. 2015 Oct;73(10):661-74. doi: 10.1093/nutrit/nuv041. Epub 2015 Sep 15. PMID 26374764
- [Background] Wang P, Tadeo X, Chew HSJ, Sapanel Y, Ong YH, Leung NYT, Chow EK, Ho D. N-of-1 health optimization: Digital monitoring of biomarker dynamics to gamify adherence to metabolic switching. PNAS Nexus. 2024 May 30;3(6):pgae214. doi: 10.1093/pnasnexus/pgae214. eCollection 2024 Jun. PMID 38881838